CLINICAL TRIAL: NCT05489289
Title: A Randomized, Double-blind, Phase III Clinical Study on the Efficacy and Safety of AK104 Versus Placebo as Adjuvant Therapy for Hepatocellular Carcinoma With High Risk of Recurrence After Curative Resection
Brief Title: A Phase III Study of AK104 as Adjuvant Therapy in HCC With High Risk of Recurrence After Curative Resection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK104-306
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK104 (Active Comparator): AK104 IV every three weeks
  Interventions: Biological: AK104
- placebo (Placebo Comparator): Placebo IV every three weeks
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: AK104 — Subjects will receive AK104 until disease progression or for a maximum of 16 cycles
  Arms: AK104
Biological: placebo — Subjects will receive placebo until disease progression or for a maximum of 16 cycles
  Arms: placebo

SUMMARY:
The efficacy and safety of AK104 as adjuvant therapy in hepatocellular carcinoma of high recurrence risk after curative resection.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of HCC without any metastasis;
2. Receiving radical resection as the only anti-tumor treatment;
3. No evidence of residual cancer found during or after the operation;
4. Presence of any high risk factor of postoperative recurrence;
5. Child-Pugh grade: A;
6. ECOG score: 0;
7. Controlled underlying causes of HCC.

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma, etc;
2. Any anti-tumor treatment other than radical surgery before randomization;
3. Precarious liver function indicated by severe complications;
4. Recent procedures or medications leading to high risk of bleeding;
5. Poorly controlled or symptomatic hypertension, congestive heart failure, arrhythmia, etc;
6. Failure of performing enhanced CT or MRI scans of the liver;
7. Recent severe infections or systemic antibiotics use;
8. Active autoimmune diseases;
9. History of other incurable malignant tumors;
10. History of transplantation;
11. Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2026-01-28 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) by BICR | Up to 48 months
  The time comfirmed by BICR from randomization to recurrence or death.

SECONDARY OUTCOMES:
12-months recurrence free survival (RFS-12) | 12 months
  The proportion of patients without recurrence or death at 12 month.
24-months recurrence free survival (RFS-24) | 24 months
  The proportion of patients without recurrence or death at 24 month.
Time to recurrence (TTR) | Up to 48 months
  The time from randomization to recurrence.
Overall survival (OS) | Up to 48 months
  The time from randomization to death for any reason.
Types and proportions of adverse events (AEs) | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No